CLINICAL TRIAL: NCT02427672
Title: The Effect of Transcranial Direct Current Stimulation of the Prefrontal Cortex on Antisocial and Aggressive Behavior
Brief Title: The Effect of Prefrontal Cortex Stimulation on Antisocial and Aggressive Behavior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 821313
Record Dates: First submitted 2015-03-26; First posted 2015-04-28 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Antisocial Behavior; Aggression
Keywords: antisocial behavior; aggression; transcranial direct current stimulation; dorsolateral prefrontal cortex; associated risk factors
MeSH Terms: conditions — Antisocial Personality Disorder; Aggression | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anodal stimulation (Experimental): Participants in the active stimulation group will undergo anodal bilateral transcranial direct current stimulation (tDCS) of the dorsolateral prefrontal cortex. tDCS will be delivered by a battery-driven, constant-current stimulator connected to three saline-soaked surface sponge electrodes. Two anodal electrodes (25cm2) will be placed over the dorsolateral prefrontal cortex bilaterally and one cathodal electrode (35cm2) will be placed at the back of the neck. Scalp electrodes will be positioned over the F3 and F4 according to the 10-20 EEG international system. A current of 1mA will be applied for 20 minutes and the current will be ramped up and down at the beginning and end of the stimulation period.
  Interventions: Device: Transcranial direct current stimulation
- Sham stimulation (Sham Comparator): The sham transcranial direct current stimulation condition will involve the same placement of the electrodes, current intensity, and ramp time as the real tDCS condition, but stimulation will only last for 30 seconds.
  Interventions: Device: Sham transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation
  Arms: Anodal stimulation
Device: Sham transcranial direct current stimulation
  Arms: Sham stimulation

SUMMARY:
This study investigates the effect of upregulating prefrontal cortex activity on antisocial and aggressive behavior and risk factors for such behavior. In the double-blind, randomized controlled trial, participants will undergo anodal transcranial direct current stimulation bilaterally to the dorsolateral prefrontal cortex or a sham stimulation. During and after stimulation, they will complete survey and laboratory measures assessing antisocial and aggressive behavior and risk factors for antisocial and aggressive behavior. Heart rate and skin conductance will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years of age
* Able to understand the nature of the study and give informed consent

Exclusion Criteria:

* History of or active neurologic, cardiovascular, or psychiatric disease
* Currently consuming anti-convulsant, anti-psychotic, or sedative/hypnotic medications
* Currently consuming anti-depressants
* History of seizures
* Metallic implants on the scalp
* Participation in other transcranial magnetic stimulation (TMS) or tDCS experiments on the same day
* History of adverse reactions to tDCS

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2015-03; Primary Completion 2017-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Raine, DPhil, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Choy O, Raine A, Hamilton RH. Stimulation of the Prefrontal Cortex Reduces Intentions to Commit Aggression: A Randomized, Double-Blind, Placebo-Controlled, Stratified, Parallel-Group Trial. J Neurosci. 2018 Jul 18;38(29):6505-6512. doi: 10.1523/JNEUROSCI.3317-17.2018. Epub 2018 Jul 2. PMID 29967006

RESULTS

PARTICIPANT FLOW:
Groups:
- Anodal Stimulation: Participants in the active stimulation group will undergo anodal bilateral transcranial direct current stimulation (tDCS) of the dorsolateral prefrontal cortex. tDCS will be delivered by a battery-driven, constant-current stimulator connected to three saline-soaked surface sponge electrodes. Two anodal electrodes (25cm2) will be placed over the dorsolateral prefrontal cortex bilaterally and one cathodal electrode (35cm2) will be placed at the back of the neck. Scalp electrodes will be positioned over the F3 and F4 according to the 10-20 EEG international system. A current of 1mA will be applied for 20 minutes and the current will be ramped up and down at the beginning and end of the stimulation period.
  Transcranial direct current stimulation
- Sham Stimulation: The sham transcranial direct current stimulation condition will involve the same placement of the electrodes, current intensity, and ramp time as the real tDCS condition, but stimulation will only last for 30 seconds.
  Sham transcranial direct current stimulation
Period: Overall Study
Arm/Group | Anodal Stimulation | Sham Stimulation
Started | 40 | 44
Completed | 39 | 42
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anodal Stimulation | Sham Stimulation | Total
Number analyzed (Participants) | 39 | 42 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.26 (4.13) | 20.17 (2.36) | 20.21 (3.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 21 | 45
  Male | 15 | 21 | 36
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 17 | 19 | 36
  Non-Caucasian | 22 | 23 | 45
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 39 | 42 | 81

OUTCOME MEASURES:

1. Primary Outcome: Change in Antisocial Behavior Inclinations at 24 Hours
Description: This will be assessed using hypothetical scenarios in which someone commits a criminal or antisocial act. The two brief scenarios describe a physical assault and a sexual assault. Participants will respond to the likelihood that they would commit the act in the scenario according to a 10-point Likert scale. Responses were measured on a scale ranging from zero (no chance at all) to ten (100 percent chance). Scores for both scenarios were summed to obtain an overall measure of intentions to commit aggression. Possible scores range from 0 to 20. A higher value indicates a greater inclination to engage in the antisocial act.
Time Frame: Baseline (an average of 15 minutes before receiving tDCS or sham) and on average, 24 hours following stimulation or sham
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Anodal Stimulation | Sham Stimulation
Number analyzed (Participants) | 39 | 42
score on a scale | 1.41 (.33) | 3.05 (.68)

2. Primary Outcome: Number of Pins Inserted Into a Virtual Voodoo Doll at 24 Hours
Description: The number of pins (between 0 and 51) that participants decide to insert into a picture of a voodoo doll on a computer that represents either a romantic partner or close friend will be recorded on average 24 hours after receiving tDCS or sham stimulation.
Time Frame: On average, 24 hours after the tDCS or sham session
Measure: Mean (Standard Error); unit: pins
Arm/Group | Anodal Stimulation | Sham Stimulation
Number analyzed (Participants) | 39 | 42
pins | 5.31 (1.90) | 2.62 (1.32)

ADVERSE EVENTS:
Time Frame: The presence of an adverse event was assessed during the course of one experimental session, from the 20-minute stimulation or sham period to the time that participants completed all study tasks, up to 1 hour.
Description: Subjects responded to a questionnaire regarding 8 possible sensations that may have resulted from tDCS.
Arm/Group | Anodal Stimulation | Sham Stimulation
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/42
Other Adverse Events (participants affected / at risk) | 39/39 | 39/42
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anodal Stimulation (N=39) | Sham Stimulation (N=42)
Itchiness (Skin and subcutaneous tissue disorders) | 36 (36) | 33 (33)
Lightheadedness (General disorders) | 19 (19) | 14 (14)
Pain (General disorders) | 20 (20) | 18 (18)
Burning (Skin and subcutaneous tissue disorders) | 23 (23) | 17 (17)
Warmth (Skin and subcutaneous tissue disorders) | 22 (22) | 19 (19)
Pinching (Skin and subcutaneous tissue disorders) | 18 (18) | 19 (19)
Iron taste (General disorders) | 4 (4) | 2 (2)
Fatigue (General disorders) | 15 (15) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-06): https://cdn.clinicaltrials.gov/large-docs/72/NCT02427672/Prot_SAP_000.pdf